CLINICAL TRIAL: NCT01591902
Title: A Prospective, Randomized, Placebo-controlled, Double-blind Clinical Trial to Evaluate Whether EGRIFTA® (Tesamorelin for Injection), 2 mg Once Daily SC, Increases the Risk of Development or Progression of Diabetic Retinopathy When Administered to HIV-infected Subjects With Abdominal Lipohypertrophy and Concomitant Diabetes
Brief Title: Diabetic Retinopathy in HIV Subjects Treated With EGRIFTA®
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Theratechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMR200147-500
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Retinopathy; HIV
MeSH Terms: conditions — Diabetic Retinopathy | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGRIFTA Treatment Grop (Experimental): Sterile, lyophilized, nonpyrogenic powder containing tesamorelin acetate with mannitol as excipient
  Interventions: Drug: Tesamorelin
- Placebo (Placebo Comparator): Placebo-controlled
  Interventions: Drug: Placebo-Control

INTERVENTIONS:
Drug: Tesamorelin — Daily 2 mg subcutaneous injections of tesamorelin
  Arms: EGRIFTA Treatment Grop
Drug: Placebo-Control — 3.0 mL vials
  Arms: Placebo

SUMMARY:
To show the non-inferiority of EGRIFTA® vs. placebo in the development or progression of Diabetic Retinopathy in HIV-infected subjects with concomitant abdominal lipohypertrophy and Type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
To date, EGRIFTA® has not been studied for longer than 1 year in human subjects, nor has EGRIFTA® been studied in Type 2 diabetic HIV-infected subjects who are receiving oral hypoglycemic agents, GLP-1 analogues, or insulin. The present study will assess the potential of EGRIFTA® to induce or exacerbate DR in HIV-infected subjects on antiretroviral therapy who have concomitant abdominal lipohypertrophy and T2DM, and explore the long-term effects of EGRIFTA® on glycemic control and major adverse cardiovascular event (MACE) in this population.

ELIGIBILITY:
Inclusion criteria:

1. Subject has given written informed consent and is willing to comply with the requirements of the protocol;
2. Subject is an adult man or woman (≥ 18 years old);
3. Subject has laboratory confirmed HIV infection;
4. Subject is receiving ART that has been stable for at least 8 weeks prior to screening;
5. Subject has physical evidence of abdominal lipohypertrophy, as determined by the examining study physician;
6. Subject has T2DM as determined by previous HbA1c ≥ 6.5%, previous fasting plasma glucose

   * ≥ 126 mg/dL (7.0 mmol/L), and/or previous 2-hour plasma glucose ≥ 200 mg/dL (11.1 mmol/L) during oral glucose tolerance testing (OGTT), and/or previous random plasma glucose ≥ 200 mg/dL (11.1 mmol/L) with symptoms of uncontrolled DM;
   * if subject has been diagnosed with T2DM and is on glucose lowering medications for greater than 1 year the above glucose parameters do not apply;
7. Subject, at the time of screening, has HbA1c between 6.0% and 12.0%;
8. Subject's diabetes has been treated for at least 1 year by diet alone, individuals who are on a stable dose (at least 3 months) of insulin, an OHA, or a GLP-1 analogue plus insulin to control diabetes are permitted if their HbA1C is below 6.0%. OHA, GLP-1 analogue, or OHA/GLP-1 analogue plus insulin according to current American Diabetes Association (ADA) guidelines, and doses have been stable for at least 3 months;
9. If the subject is using lipid lowering drugs, the dose must be stable for at least 2 months prior to screening;
10. Subject must have an electrocardiogram (ECG) without clinically significant abnormalities within 6 months prior to screening;
11. Pre-menopausal women of childbearing potential are eligible only if they are not pregnant (negative urine pregnancy tests at screening and baseline) or lactating and are using an acceptable form of birth control prior to study entry and for at least 2 months after completing treatment. Acceptable contraception is defined as two barrier methods, or one barrier method with a spermicide, or an intrauterine device, or an oral contraceptive;
12. Women of non-childbearing potential must be post-menopausal (no menses for more than 1 year) or surgically sterile (tubal ligation or hysterectomy);
13. Women over 40 years old must have a negative mammogram within 6 months prior to screening or a mammogram will be taken at screening;
14. Men must have a normal prostate exam and a prostate specific antigen (PSA) Individuals who are on a stable dose (at least 3 months) of insulin, less than or equal to 5 ng/mL within 6 months prior to screening or PSA and, for men 50 years of age or older, a prostate specific antigen will be measured at screening

Exclusion Criteria:

1. Subject has Type 1 DM;
2. Subject has body mass index (BMI) < 18.5 kg.m2;
3. Subject has or has had an opportunistic infection or acquired immune deficiency syndrome (AIDS)-defining illness within 3 months of screening;
4. Subject has or has had a malignancy or, for women, personal or family (first degree relative) history of breast cancer. Exceptions are basal cell carcinoma, in situ carcinoma of the cervix, in situ anal carcinoma, treated and stable cutaneous squamous cell carcinoma. and stable Kaposi's sarcoma;
5. Pre-existing PDR or severe non-PDR (NPDR), defined as an ETDRS level of ≥ 53 in either eye;
6. Subject has or has had cytomegalovirus (CMV) retinitis, toxoplasmosis, or any other ocular infection that would prevent evaluation of DR;
7. Subject has previously been treated for DR (treatments such as laser photocoagulation, intravitreal injection, or vitrectomy);
8. Subject has any of the following illnesses or conditions:

   1. hypopituitarism, history of pituitary tumor or pituitary surgery;
   2. untreated hypothyroidism;
   3. head irradiation or head trauma that has affected the somatotropic axis;
   4. uncontrolled hypertension, defined as systolic pressure > 140 mm Hg and diastolic pressure > 90 mm Hg;
   5. unstable CV condition, defined as:

   i. acute MI; ii. unstable angina; iii. decompensated congestive heart failure (CHF, new onset or exacerbation); iv. stroke; v. history of any of the above within 6 months prior to screening; f. hepatic abnormality, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal (3 x ULN); g. renal abnormality, defined as serum creatinine > 2 x ULN; h. lipid metabolism abnormality, defined as fasting triglycerides > 1500 mg/dL; i. anemia, defined as hemoglobin ≤ 7 g/dL;
9. Drug or hormone use as follows

   1. Men: change in regimen or supraphysiological dose of testosterone within 2 months prior to screening;
   2. anabolic steroids, GH, GH secretagogue, GHRF products or analogs (including EGRIFTA®), IGF-1, or IGF binding protein 3 (IGFBP 3) within 6 months prior to screening;
10. Drug or alcohol dependence within 6 months prior to screening;
11. Subject is using or has used anorectics, anorexigenics, or anti-obesity agents within 3 months prior to screening;
12. Subject is pregnant or nursing;
13. Other significant disease that, in the Investigator's opinion, would exclude the subject from the trial;
14. Participation, within 30 days prior to screening, in another clinical trial of an investigational agent that could affect IGF-1 levels;
15. Known hypersensitivity to the study drug treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Difference in percentages of subjects with a 3-step or greater progression (from both eyes) on the Early Treatment Diabetic Retinopathy Study (ETDRS) PERSON scale. | 3 years
  Subjects will undergo an opthamologic examination including fundus photographs at 3 month intervals for duration of 36 months

SECONDARY OUTCOMES:
Change from baseline in HbA1c by intensification of concomitant diabetic treatment | 3 years
  HbA1c values will be obtained at screening at month 3, 6, 12, 18, 24, 30 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn De Chantal
Locations (24):
- United States (24):
  - Southwest Center for HIV/AIDS, Phoenix, Arizona
  - Spectrum Medical Group, Phoenix, Arizona
  - 5P21 Rand Schrader Clinic, Los Angeles, California
  - University of California CARE Clinic, Los Angeles, Los Angeles, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - UCSD Antiviral Research Center, San Diego, California
  - VAMC, Infectious Disease Section 111W, San Francisco, California
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Gary J. Richmond, M.D., PA, Fort Lauderdale, Florida
  - Orange County Health Department, Orlando, Florida
  - Triple O Research Institute, West Palm Beach, Florida
  - Rowan Tree Medical , P.A., Wilton Manors, Florida
  - Be Well Medical Center, P.C., Berkley, Michigan
  - Southampton Clinical Research, Inc d.b.a. Central West Clinical Research, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Harold Hamm Diabetes Center at the University of Oklahoma, Oklahoma City, Oklahoma
  - Fanno Creek Clinic, LLC, Portland, Oregon
  - Central Texas Clinical Research, Austin, Texas
  - St. Hope Foundation, Inc., Bellaire, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Atten: HIV Research Unit, Dallas, Texas
  - Research Access Network, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington